CLINICAL TRIAL: NCT03845439
Title: Estimate of the Time Since Death Based on the Post Mortem Quantification of the Tau Protein in the Cerebrospinal Fluid
Brief Title: Estimate of the TSD Based on the Quantification of the Tau Protein in CSF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0369-Uf5003
Record Dates: First submitted 2019-02-18; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Time of Death
Keywords: tau; post mortem interval; cerebrospinal fluid; immunoassay; biomarker; forensic medicine
MeSH Terms: conditions — Pick Disease of the Brain | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Lumbar puncture — Lumbar puncture

SUMMARY:
Background: The accurate estimation of the time of death is a challenge in forensic medicine, as the methods routinely used to assess the post-mortem interval (PMI) are far from being precise. Recent developments in biochemical techniques may provide the opportunity to assist in more precise estimation of the time of death. The focus has been placed on the study of the biochemical profiles of closed compartment body fluids, as they are longer preserved than blood after death and subject to confined post-mortem chemical changes. Cerebrospinal fluid (CSF) has been considered as a suitable fluid to investigate these changes, as it is easy to sample and found in large amount.

Due to its closeness to the central nervous system (CNS), CSF is used in clinical settings for the diagnosis of various CNS disorders such as Alzheimer's disease, whose diagnosis is mainly based on the increase of the concentrations of Tau protein and its phosphorylated isoform (p-Tau) in CSF. A post mortem leakage of Tau into the CSF has also been shown, reflecting progressive neuronal death as in Alzheimer's disease. In this exploratory, cross-sectional study, we investigated Tau in post mortem CSF as a potential biomarker of the time of death.

Objectives: The main objective was to assess the correlation between the concentration of Tau in CSF and the PMI. The secondary objectives were (1) to determine the inter-individual variability of the concentration of Tau for a same PMI; (2) to determine the kinetics of this concentration over time in the same individual; (3) to determine the variability of this concentration according to the site of collection (lumbar vs. sub-occipital).

DETAILED DESCRIPTION:
Background: The accurate estimation of the time of death is a challenge in forensic medicine, as the methods routinely used to assess the post-mortem interval (PMI) are far from being precise. Recent developments in biochemical techniques may provide the opportunity to assist in more precise estimation of the time of death. The focus has been placed on the study of the biochemical profiles of closed compartment body fluids, as they are longer preserved than blood after death and subject to confined post-mortem chemical changes. Cerebrospinal fluid (CSF) has been considered as a suitable fluid to investigate these changes, as it is easy to sample and found in large amount.

Due to its closeness to the central nervous system (CNS), CSF is used in clinical settings for the diagnosis of various CNS disorders such as Alzheimer's disease, whose diagnosis is mainly based on the increase of the concentrations of Tau protein and its phosphorylated isoform (p-Tau) in CSF. A post mortem leakage of Tau into the CSF has also been shown, reflecting progressive neuronal death as in Alzheimer's disease. In this exploratory, cross-sectional study, we investigated Tau in post mortem CSF as a potential biomarker of the time of death.

Objectives: The main objective was to assess the correlation between the concentration of Tau in CSF and the PMI. The secondary objectives were (1) to determine the inter-individual variability of the concentration of Tau for a same PMI; (2) to determine the kinetics of this concentration over time in the same individual; (3) to determine the variability of this concentration according to the site of collection (lumbar vs. sub-occipital).

Materials and methods: The study was reviewed and approved by the Ethics Committee of the University Hospital of Montpellier. Post mortem CSF samples were collected from 80 adult cadavers whose time of death was precisely known, at the mortuary of the University Hospital of Montpellier. Individuals with neurological disorders and head trauma were excluded from the study, as well as subjects with unknown past medical history or cause of death. CSF samples were removed by cisternal and lumbar punctures at the time of arrival at the mortuary, before refrigeration. A few mL of CSF were obtained at each tap in clean, sterile polypropylene tubes, using a 18G lumbar puncture needle. The cadavers were divided into four groups according to the PMI (n=25 in each group). The samples were taken 0-6 h (group A), 6-12 h (group B), 12-18 h (group C) and 18-24 h (group D) after death. Additionally, CSF samples were collected every 3h from 10 cadavers during the first 15 h post mortem. All cadavers were kept at room temperature (+20 ± 2°C) during sample collection. CSF samples were transferred at +4°C to the laboratory where they were centrifuged for 10 min (+4°C, 1000 g). The clear supernatant was divided into aliquots then stored at -80°C until analysis. The rectal and tympanic temperatures were measured at the time of CSF collection using a probe thermometer.

Concentrations of Tau and and its phosphorylated isoform (p-Tau) were measured by conventional immunoassays, while total protein concentration was determined using a bicinchoninic acid protein assay.

The correlation coefficient between the concentration of Tau in CSF and the PMI was calculated in each case. The inter-individual variability was assessed by measuring the standard deviation (SD) of the mean concentration of Tau in each group. Linear regression analysis (adjusted for confounders) was used in assessing whether Tau concentration was dependent on the PMI. Paired Student's t-test was used to assess the variability of Tau concentration depending on the site of CSF collection

ELIGIBILITY:
Inclusion criteria:

- Adult cadavers whose time of death is precisely known

Exclusion criteria:

- Individuals with neurological disorders, head trauma or with unknown past medical history or cause of death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient undergoing a forensic autopsy
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Tau concentration in CSF | 1 day
  Tau concentration in CSF

SECONDARY OUTCOMES:
pTau concentration in CSF | 1 day
  pTau concentration in CSF

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Antoine PEYRON, MD, Study Director — University Hospital, Montpellier
Locations (1):
- PEYRON, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided